CLINICAL TRIAL: NCT06757712
Title: Nonlinear Versus Linear Periodized Resistance Training on Quality of Life in Females With Hypothyroidism
Brief Title: Periodization Resistance Training on Quality of Life in Females With Hypothyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mahmoud Mohamed Abd elhady, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005442
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non linear periodization exercise + medical treatment (Experimental): It will consist of 25 females, who will receive non linear periodization exercise in addition to their medical treatment.
  Interventions: Other: non linear periodization exercise; Drug: medical treatment
- linear periodization exercise + medical treatment (Experimental): It will consist of 25 females, who will receive linear periodization exercise in addition to their medical treatment.
  Interventions: Other: linear periodization exercise; Drug: medical treatment
- medical treatment (Active Comparator): It will consist of 25 females, who will receive their medical treatment only.
  Interventions: Drug: medical treatment

INTERVENTIONS:
Other: non linear periodization exercise — The non-linear periodized resistance training program follows a 12-week schedule with varying intensity levels across three training days per week. The intensity fluctuates between very light (VL), light (L), moderate (M), heavy (H), and very heavy (VH) workouts, distributed strategically throughout the week. Each training day implements different intensity levels, and an active rest day follows any workout session.
  Arms: non linear periodization exercise + medical treatment
Other: linear periodization exercise — The linear periodization exercise program spans 12 weeks with systematically varied training parameters. During weeks 1-2, participants perform 3 sets of 10 repetitions, followed by 3 sets of 8 repetitions in weeks 3-4. The program progresses to 4 sets of 6 repetitions in weeks 5-6, then 3 sets of 6 repetitions during weeks 7-8. The final phases consist of 4 sets of 4 repetitions in weeks 9-10, concluding with 3 sets of 4 repetitions in weeks 11-12. Training loads advance through autoregulatory progression, where participants progress at their individual pace under supervision. While sets and repetitions remain fixed within each phase, load progression is determined by performance in the final set of each exercise, ensuring safe and effective advancement.
  Arms: linear periodization exercise + medical treatment
Drug: medical treatment — The medical treatment will be received for 12 weeks.

SUMMARY:
This study will be conducted to compare between the effect of nonlinear and linear periodized training on quality of life in females with hypothyroidism.

DETAILED DESCRIPTION:
Worldwide, the incidence of individuals with thyroid dysfunction is increasing and represents approximately 30-40% of the patients seen in an endocrine clinic; thus, it is one of the leading endocrine disorders.The undiagnosed thyroid dysfunction especially subclinical and clinical hypothyroidism may increase cardiovascular risk factors.

The prevalence of hypothyroidism depends on many factors, such as age, sex and geographical factors. It's also a diet related disorder and it's usually seen when the daily intake of iodine falls below 25μg.

Hypothyroidism tends to affect women more often than men and can manifest at any age, typically observed between 40 and 70 years. No specific racial predilection has been identified in studies regarding this condition. regular exercise can improve quality of life in patients with subclinical hypothyroidism by increasing physical activity level/fitness and reducing the signs and symptoms of the disease. Exercise may therefore potentiate the effectiveness of levothyroxine and help hypothyroid individuals improve their quality of life.

Periodization of resistance training or planned changes in training volume and intensity are used to maximize strength and fitness gains. The most common of periodized resistance training plans is linear also termed classic or strength/power periodization and nonlinear periodization. The biggest difference between these two types of training plans is with nonlinear periodization changes in training volume and intensity are made more frequently. The most common type of nonlinear periodization is daily nonlinear periodization where substantial changes in training intensity and volume are made from one training session to the next training session.

So, this study will be conducted to compare between the effect of non linear and linear periodized resistance training on quality of life in females with hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Be controlled hypothyroidism (TSH level within 0.5 - 4.5 mU/L)
* Be ranged from 35 to 45 years
* Female patients
* Body Mass Index 30-34.9 kg/m2 .
* triglyceride-glucose (TyG) index > 4.5

Exclusion Criteria:

* history of pulmonary disease
* Patients with uncontrolled coronary or cerebrovascular disease
* Those who underwent musculoskeletal surgery within the previous year
* Recent history of lower and upper limb fracture , hip and shoulder dislocation.
* Cognitive impaired patients
* Patients with history of epilepsy
* Patients who participating in any other exercise program

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Serum thyroid stimulating hormone (TSH) level | 12 weeks
  It will be measured by ELISA kits. This kit is an Enzyme Linked Immunosorbent Assay (ELISA). (Precheck bio, inc, @ EIA KIT, USA).
FreeT4 (thyroxine) level | 12 weeks
  It will be measured by ELISA kits. This kit is an Enzyme Linked Immunosorbent Assay (ELISA). (Precheck bio, inc, @ EIA KIT, USA).
Health related Quality of life questionnaire | 12 weeks
  The Health related Quality of life will be assessed using short form 12 (SF-12), which uses only 12 questions to measure functional health and well being from the patient's perspective. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

SECONDARY OUTCOMES:
Triglyceride-glucose (TyG) index | 12 weeks
  The triglyceride-glucose (TyG) index indirectly assesses insulin resistance through a mathematical model that uses only laboratory data on fasting plasma triglyceride and glucose concentrations. The TyG index will be calculated according to the formula: fasting triglycerides (mg/dL) × fasting plasma glucose (mg/dL) /2].
Hand grip strength | 12 weeks
  It will be measured before and after treatment using a hand-held dynamometer (HHD), which offers a reliable and valid method.
9-item Fatigue Severity Scale (FSS) | 12 weeks
  It will be used before and after treatment to assess fatigue severity. The FFS is a nine-item unidimensional questionnaire scored on a seven-point Likert scale, with high sum scores indicating greater fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Gharib Mohamed Elnahas, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Suez University, Suez, Egypt